CLINICAL TRIAL: NCT01566877
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose, Dose-Escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of AVI-7288 in Healthy Adult Volunteers
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of AVI-7288 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7288-us-101; W9113M-10-C-0056 (Other Grant/Funding Number: Transformational Medical Technologies, US Dept. of Defense)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Marburg Hemorrhagic Fever
Keywords: Multiple Ascending Dose (MAD); Marburg Virus; Post Exposure Prophylaxis
MeSH Terms: conditions — Marburg Virus Disease | interventions — AVI-7288; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AVI-7288 (Active Comparator): AVI-7288 is a phosphorodiamidate morpholino oligomer with positive charges (PMOplus™) that targets Marburg virus nucleoprotein (NP). AVI-7288 is supplied in 5 mL vials containing 5 mL AVI-7288 at a concentration of 50 mg/mL. The dose levels of AVI-7288 will vary in four cohort's.
  Interventions: Drug: AVI-7288
- Placebo (Placebo Comparator): Placebo control consists of approximately 150 mL normal saline solution administered by IV infusion over 30 minutes once a day for 14 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AVI-7288 — Cohort 1: AVI-7288 at 1 mg/kg IV; Cohort 2: AVI-7288 at 4 mg/kg IV;Cohort 3: AVI-7288 at 8 mg/kg IV; Cohort 4: AVI-7288 at 12 mg/kg IV
  The amount of AVI-7288 required to administer the required dose will be diluted to a volume of approximately 150 mL with normal saline solution (NSS) and given by IV infusion over 30 minutes once a day for 14 days. Infusions will be administered at approximately the same time each day.
  Arms: AVI-7288
Other: Placebo — Normal Saline Solution (NSS)
  Other Names: Normal Saline Solution (NSS)
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of healthy male and female subjects with intravenous (IV) infusions of AVI 7288 compared to matched placebo in and to evaluate the pharmacokinetics (PK).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and tolerability of 14 once daily intravenous (IV) infusions of ascending doses of AVI 7288 compared to matched placebo in healthy male and female subjects.

To evaluate the pharmacokinetics (PK) of 14 once daily doses of AVI-7288 in healthy male and female subjects

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all of the following criteria to be eligible for this study.

1.Man or woman 18 to 50 years of age, inclusive, at the time of screening. 2.Body mass index 18 kg/m2 to 35 kg/m2, inclusive, at the time of screening and Check-in (Day -1).3.Good general health (no chronic health conditions) as determined by the Investigator.4.Female subjects must be of non-childbearing potential or must, in conjunction with their sexual partner(s), use 2 forms of medically acceptable barrier contraception (e.g., a diaphragm with spermicidal jelly in conjunction with a male condom) during the screening period and for the entire duration of the study including the 28-day post last dose follow-up.5.Male subjects must either be sterile or agree to use, for the entire duration of the study and for 90 days post last dose follow-up, a male condom and the female sexual partner must also use a medically acceptable form of birth control (e.g. oral contraceptives). 6. Male subjects must agree not to donate sperm for at least 90 days after the last infusion of study medication. 7.Able to understand the requirements of the study, to provide written informed consent (as evidenced by signature on an informed consent document that is approved by an Institutional Review Board (IRB), and agree to abide by the study restrictions.

Exclusion Criteria:

A subject who meets any of the following criteria will be excluded from this study.

1.Pregnancy or breastfeeding. 2. A positive urine or blood screen for drugs of abuse, including alcohol. 3.Use of any tobacco- or nicotine-containing products(including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to Check-in (Day -1). 4.Donated blood within 90 days or plasma within 30 days of first dose on Day 1. 5.A positive cotinine test indicating recent nicotine use.6.Active substance abuse or any medical or psychiatric condition that could jeopardize the subject's safety or the subject's ability to comply with the protocol. 7.Use of any medications apart from vitamins, acetaminophen or hormonal contraception within 14 days of first dose on Day 1. Subjects with mild seasonal allergies may use antihistamines at the discretion of the Investigator after discussion with the Sponsor Medical Monitor.8.Participation in any interventional clinical trial within 45 days of first dose on Day 1 (i.e., received any other investigational drug).9. Recipient of an organ transplant (solid or hematopoietic). 10.Prolonged QTcF interval >(440 ms) for males or > 460 ms for females using the average of the triplicate ECGs collected during screening, on Day -1, or just prior to dosing on Day 1. 11.Other clinically significant electrocardiogram (ECG) abnormality, as determined by the Investigator. 12.Any clinically significant abnormal hematology, chemistry, coagulation, or urinalysis value, as determined by the Investigator. 13.Glomerular filtration rate (GFR) of < 90 mL/min, based on the Modification of Diet in Renal Disease equation.14.Urine-albumin-to-creatinine ratio (UACR) > 30 mg/g. 15.Positive test for human immunodeficiency virus (HIV-1 serology) or known HIV infection. 16.Positive result for hepatitis B surface antigen (HBsAg) or for hepatitis C virus (HCV) antibody.17.Use of alcohol-containing foods or beverages within 72 hours prior to Check-in on Day -1.18.Use of caffeine-containing foods or beverages within 24 hours prior to Check-in on Day 1. 19.Febrile illness or significant infection within 48 hours before administration of the first dose of study drug on Day 1.

Note: Inclusion of each subject will be reviewed with a member of Sarepta Therapeutics Clinical Personnel prior to enrollment in the trial. Written approval from a member of Sarepta Therapeutics Clinical Personnel is required prior to randomization.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The outcome measure is safety, as assessed through adverse event evaluation and serial clinical assessments. | daily during dosing period with follow up on Day 21 and Day 42

SECONDARY OUTCOMES:
The outcome measures are Serial PK Day 1 over 24 hours(predose, 10minutes post, 30 minutes post, 1 hour 1.5, 2, 4, 6,. 8, 12,16,24 hours post dose), daily trough level and on Day 14 (last day of dosing) serial PK until 48 hours post last dose. | 2 Weeks
  Efficacy will not be assessed in a Phase I study.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Al-Ibrahim, MD, Principal Investigator — SNBL
Locations (1):
- SNBL Clinical Pharmacology Center, Inc., Baltimore, Maryland, United States

REFERENCES:
- [Derived] Heald AE, Charleston JS, Iversen PL, Warren TK, Saoud JB, Al-Ibrahim M, Wells J, Warfield KL, Swenson DL, Welch LS, Sazani P, Wong M, Berry D, Kaye EM, Bavari S. AVI-7288 for Marburg Virus in Nonhuman Primates and Humans. N Engl J Med. 2015 Jul 23;373(4):339-48. doi: 10.1056/NEJMoa1410345. PMID 26200980